CLINICAL TRIAL: NCT03814382
Title: Exploring the Use of Acupuncture to Reduce Agitation, Irritability and Anxiety in Alzheimer's Disease and Alzheimer's Disease Related Dementias Utilizing Noninvasive Measures of Autonomic Nervous System Physiology and Actigraphy Biomarkers
Brief Title: Acupuncture to Reduce Anxiety in Alzheimer's Disease (AD) and AD Related Dementias
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination of study funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven E Arnold, Managing Director Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018P002480
Record Dates: First submitted 2018-12-19; First posted 2019-01-24 (Actual); Results first posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Alzheimer's Dementia With Behavioral Disturbance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Acupuncture (Experimental): All subjects will receive up to 10 needles for 20 minutes for 1 treatment using acupuncture needles.
  Interventions: Device: Acupuncture needle

INTERVENTIONS:
Device: Acupuncture needle — Acupuncture needle

SUMMARY:
The purpose of this study is to investigate the influence of acupuncture on heart rate variability, skin conductance (sweating), and rated behavioral expression of agitation, irritability, and anxiety and mood in qualifying adults with a diagnosis of cognitively unimpaired, or probable Alzheimer's Disease, Frontotemporal Dementia or Dementia with Lewy Bodies. Study subjects will all receive one real acupuncture treatment; mood scales will be assessed before and after.

Massachusetts General Hospital is paying for this research to be done.

DETAILED DESCRIPTION:
Acupuncture is a system of integrative medicine that involves pricking the skin or tissues with needles, used to alleviate pain and to treat various physical, mental, and emotional conditions. Originating in ancient China, acupuncture is now widely practiced globally.

ELIGIBILITY:
Inclusion Criteria:

* Ages 55-95 inclusive, male or female.
* Diagnosis of CU, or probable AD, FTD or DLB as determined by established clinical criteria at screening14.
* For the AIA symptomatic groups, a score of > 2 for Severity on at least 1 of the AIA-relevant items on the NPI-Q, i.e., Anxiety, Irritability/Lability, Agitation or Aggression.
* For the CU and no neuropsychiatric symptoms group, NPI-Q score must be 0 for AIA-relevant items, i.e., Anxiety, Irritability/Lability, Agitation or Aggression.
* No concurrent use of therapies with prohibitive effects on interpretation of HRV and SC measurements, e.g., those with major direct adrenergic or anticholinergic activities.
* Stable doses (>2 weeks) of concurrent dementia or psychiatric drugs for those applicable.

Exclusion Criteria:

* Atrial or junctional arrhythmias or other cardiac conditions, including pacemakers or other implantable devices that affect RR intervals or their measurement.
* AIA symptoms or dementia so severe that subject cannot assent and cooperate with all study procedures or requires immediate rescue medication for behavioral control.
* Seizure disorders or other potentially confounding medical, neurological or longstanding psychiatric illnesses.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison McManus, Principal Investigator — MGH
Locations (1):
- Clinical Translational Research Unit, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acupuncture
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acupuncture
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.33 (7.685)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Variability as Measured by BioStamp
Description: We propose that acupuncture might acutely change Heart Rate Variability in AD/ADRD subjects with AIA. BioStamp will continuously measure participants' heart rate for 48 hours.
Time Frame: 24 hours
Population: The data was so noisy that is was unable to be analyzed
Arm/Group | Acupuncture
Number analyzed (Participants) | 0

2. Primary Outcome: Galvanic Skin Response
Description: We propose that acupuncture might acutely change Galvanic Skin Response in AD/ADRD subjects with AIA. Galvanic Skin Response measures sweating output in participants' fingers. The sweating response will be captured at both study visits.
Time Frame: 24 hours
Population: The data was so noisy that is was unable to be analyzed
Arm/Group | Acupuncture
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 48 hours
Description: AE definitions do not differ from this trial.
Arm/Group | Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
This study Investigated a wearable technology for HRV and galvanic skin response as an indicator of autonomic function for use in tracking people over time in clinical trials. We observed high day to day variability in measures that led us to conclude that this technology is not useful for our clinical trials in its current state.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT03814382/Prot_SAP_000.pdf